CLINICAL TRIAL: NCT05466123
Title: Bringing Life to Those Near Death: Assessing the Use of Virtual Reality Technology in Palliative Care
Brief Title: Bringing Life to Those Near Death
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Chimere E. Bruning, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-007346
Record Dates: First submitted 2022-07-15; First posted 2022-07-20 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual reality intervention in palliative care patients (Experimental): Palliative care patients with a limited life expectancy will participate in a virtual reality experience for 10-30 minutes
  Interventions: Behavioral: Virtual Reality

INTERVENTIONS:
Behavioral: Virtual Reality — Simulated travel destination or activity of the participants choosing that would otherwise be inaccessible

SUMMARY:
The purpose of this study is to assess whether virtual reality technology can reduce anxiety, depression, and emotional distress screening scores in palliative care patients.

ELIGIBILITY:
Inclusion Criteria;

* A terminal or end-stage condition with an expected prognosis of a year or less.
* An established palliative care patient.
* English-speaking.
* Able to wear virtual reality equipment (goggles, etc.).
* Subject or Caregiver able to provide consent.

Exclusion Criteria:

* Younger than 18 years of age.
* Lack of a prognosis of approximately 1 year or less.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in anxiety | Baseline, post-intervention approximately 30 minutes
  Measured using the self-reported Generalized Anxiety Disorder-7 (GAD-7) questionnaire. Subjects rank how often they have been bother by specific problems within the last 2 weeks on a scale of 0 being not at all and 3 being nearly every day. Total scores range from 0-20, with higher scores indicating more anxiety severity.
Change in emotional distress | Baseline, post-intervention approximately 30 minutes
  Measured using the self-reported Distress from Death and Dying Survey. Subjects rank their distress on a scale or 0-10, 0 being no distress at all, and 10 being completely distressed. Total scores range from 0-130, with higher scores indicating more distress severity.

CONTACTS AND LOCATIONS:
Overall Officials: Chimere Bruning, PA-C, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No